CLINICAL TRIAL: NCT01333904
Title: A Four-Part Study to Evaluate the Safety, Tolerability and Pharmacodynamic Effects of PUR118 and Placebo in Normal Healthy Volunteers and Subjects With COPD
Brief Title: Safety, Tolerability, and Pharmacodynamic Effect Study of PUR118
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Collaborators: Quotient Bioresearch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 601-0004
Record Dates: First submitted 2011-04-07; First posted 2011-04-12 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PUR118 (Experimental)
  Interventions: Drug: PUR118

INTERVENTIONS:
Drug: PUR118 — inhaled

SUMMARY:
The purpose of this study is to establish single and multiple dose safety in healthy subjects and subjects with mild chronic pulmonary obstructive disease (COPD). In addition, the study will evaluate preliminary proof of concept endpoints in COPD subjects such as biomarkers in sputum and mucociliary clearance.

DETAILED DESCRIPTION:
The proposed initial trial in healthy subjects and subjects with mild COPD will establish the tolerability of PUR118 in these subjects over single and short multi-day dosing periods. The study will also provide preliminary data regarding PUR118's potential impact on biomarkers in COPD. Finally, this trial will assess PUR118's effect on mucociliary clearance. This is a four part study enrolling healthy volunteers in a single ascending dose design (SAD; Part I), followed by multiple ascending dose design (MAD; Part II). Contingent on demonstration of safety in a healthy subject population, the study will enroll mild COPD subjects for a short multi-dose design (Part III) incorporating safety and pharmacodynamic endpoints. Lastly Part IV of the trial will assess the effect of PUR118 on mucociliary clearance in mild COPD subjects.

ELIGIBILITY:
Main Inclusion Criteria Parts I & II

* Healthy males or non pregnant, non lactating healthy females;
* Age 18-65 years of age;
* Must be willing and able to communicate in English and participate in the whole study;
* Must provide written informed consent.

Main Exclusion Criteria Parts I & II

* Current smokers and those who have smoked within the last 12 months;
* Females of child bearing age not willing to use an acceptable form of contraception;
* Presence or history of allergy requiring treatment;
* Serious adverse reaction or hypersensitivity to any drug;

Main Inclusion Criteria: Parts III and IV

* Males or non pregnant, non lactating females;
* Age 45-70 years;
* Current (Part III only) or ex-smokers who at least a 15 pack-year smoking history. For Part IV, subjects must be non-smokers for at least 3 months;
* Medically stable, with no evidence of uncontrolled co-existing conditions at screening;
* Must not be taking any inhaled or oral corticosteroids;
* FEV1/FVC ratio <70% and FEV1 60 - 80% (or >/= 60% for Part IV only) of predicted following administration of a bronchodilator;
* Patients must have a medical history of COPD confirmed by their General Practitioner (GP) or treating hospital physician or must have a chest x-ray (CXR) which is normal or consistent with mild COPD and excludes other clinically significant respiratory abnormalities;
* Must be willing and able to communicate in English and participate in the whole study;
* Must provide written informed consent.

Main Exclusion Criteria: Parts III and IV

* Must agree to use an adequate method of contraception;
* Upper respiratory tract infection within 30 days of the first study day, or lower respiratory tract infection within the last 60 days;
* Patients taking medication that may affect the respiratory tract within 14 days of the first study day other than their usual COPD medication;
* No active exacerbations requiring antibiotics or steroids within 60 days of dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by changes in clinical signs and symptoms, clinical safety laboratory tests, vital signs, ECG, spirometry, oxygen saturation, telemetry and adverse events | 2 weeks

SECONDARY OUTCOMES:
Assessment of biomarkers of inflammation and COPD in induced sputum in mild COPD subjects after short multi-dosing with PUR118 compared to baseline | 2 days
Assessment of changes in mucociliary clearance after treatment with PUR118 in mild COPD subjects compared to baseline | single dose

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MD, Principal Investigator — Quotient Bioresearch
Locations (1):
- Quotient Bioresearch, Nottingham, United Kingdom, United Kingdom